CLINICAL TRIAL: NCT01620489
Title: Efficacy and Safety of Liraglutide Versus Placebo as add-on to Existing Diabetes Medication in Subjects With Type 2 Diabetes and Moderate Renal Impairment. A 26-week Double-blind Placebo-controlled, Randomised, Multicentre, Multi-national, Parallel-group Trial
Brief Title: Efficacy and Safety of Liraglutide Versus Placebo as add-on to Existing Diabetes Medication in Subjects With Type 2 Diabetes and Moderate Renal Impairment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN2211-3916; 2011-002968-24 (EudraCT Number); U1111-1122-3303 (Other: WHO)
Record Dates: First submitted 2012-06-13; First posted 2012-06-15 (Estimated); Results first posted 2014-10-30 (Estimated); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lira 1.8 mg (Experimental)
  Interventions: Drug: liraglutide
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: liraglutide — 1.8 mg administered once daily subcutaneously (s.c., under the skin) as add-on to the subject's stable pre-trial oral antidiabetic drug (OAD) and/or insulin regimen.
  Arms: Lira 1.8 mg
Drug: placebo — Administered once daily subcutaneously (s.c., under the skin) as add-on to the subject's stable pre-trial oral antidiabetic drug (OAD) and/or insulin regimen.
  Arms: Placebo

SUMMARY:
This trial is conducted in Europe and the United States of America (USA). The aim of this trial is to investigate the efficacy and safety of liraglutide in subjects with type 2 diabetes and moderate renal impairment.

The trial medication will be add-on to the subject's stable pre-trial OAD and/or insulin regimen.

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed with type 2 diabetes with stable diabetes treatment (unchanged medication and unchanged dose) for 90 days prior to the screening visit including: Monotherapy or any duo-combinations of metformin and/or SUs and/or pioglitazone. Metformin should be used with caution in subjects with moderate renal failure and must be used in accordance with local metformin labelling or guidelines. Or Monotherapy or any combinations of metformin and/or pioglitazone and/or basal or premix insulin. Insulin adjustments (total daily dose) below or equal to 10% within 90 days prior to the screening visit as confirmed by the investigator are acceptable. Metformin should be used with caution in subjects with moderate renal failure and must be used in accordance with local metformin labelling or guidelines. Combination of pioglitazone and insulin should be used with caution and according to local labelling or guidelines
* HbA1c 7-10% (both inclusive)
* Moderate renal impairment diagnosed more than 90 days prior to the screening visit and confirmed by an eGFR (glomerular filtration rate) of 30-59 mL/min/1.73 m2 per MDRD (modification of diet in renal disease) formula at the screening visit
* Body Mass Index (BMI) 20-45 kg/m^2 (both inclusive)

Exclusion Criteria:

* Recurrent severe hypoglycaemia or hypoglycaemic unawareness as judged by the investigator
* Treatment with antidiabetic medication(s) other than stated in the inclusion criteria in a period of 90 days prior to screening. Previous short-term (below or equal to 7 days in total) treatment with rapid-or short-acting insulin in connection with intercurrent illness is allowed at the discretion of the investigator
* Impaired liver function, defined as ALAT (alanine aminotransferase) above or equal to 2.5 times upper normal limit
* History of chronic pancreatitis or idiopathic acute pancreatitis
* Within the past 180 days any of the following: Episode of unstable angina, acute coronary event, cerebral stroke/transient ischemic attack (TIA) or other significant cardiovascular event (including e.g. arrhythmias or conduction delays on ECG (electrocardiogram))
* Heart failure defined as New York Heart Association (NYHA) class IV
* A systolic blood pressure above or equal to 180 mmHg or a diastolic blood pressure above or equal to 100 mmHg
* Rapidly progressing renal disease (e.g., acute glomerulonephritis) at the discretion of the investigator
* Use of immunosuppressive treatment within 90 days prior to screening
* Diagnosis or treatment for cancer in the previous 5 years (except basal cell skin cancer or squamous cell skin cancer)
* Proliferative retinopathy or maculopathy requiring acute treatment as judged by the investigator

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 279 (Actual)
Dates: Start 2012-06-14 (Actual); Primary Completion 2013-08-20 (Actual); Study Completion 2013-08-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (85):
- United States (50):
  - Novo Nordisk Investigational Site, Concord, California
  - Novo Nordisk Investigational Site, La Jolla, California
  - Novo Nordisk Investigational Site, Los Angeles, California
  - Novo Nordisk Investigational Site, Monterey, California
  - Novo Nordisk Investigational Site, San Diego, California
  - Novo Nordisk Investigational Site, San Ramon, California
  - Novo Nordisk Investigational Site, Torrance, California
  - Novo Nordisk Investigational Site, Tustin, California
  - Novo Nordisk Investigational Site, Ventura, California
  - Novo Nordisk Investigational Site, Golden, Colorado
  - Novo Nordisk Investigational Site, Boynton Beach, Florida
  - Novo Nordisk Investigational Site, Jacksonville, Florida
  - Novo Nordisk Investigational Site, Miami, Florida
  - Novo Nordisk Investigational Site, Pembroke Pines, Florida
  - Novo Nordisk Investigational Site, Plantation, Florida
  - Novo Nordisk Investigational Site, St. Petersburg, Florida
  - Novo Nordisk Investigational Site, Atlanta, Georgia
  - Novo Nordisk Investigational Site, Roswell, Georgia
  - Novo Nordisk Investigational Site, Avon, Indiana
  - Novo Nordisk Investigational Site, Franklin, Indiana
  - Novo Nordisk Investigational Site, Greenfield, Indiana
  - Novo Nordisk Investigational Site, Muncie, Indiana
  - Novo Nordisk Investigational Site, Slidell, Louisiana
  - Novo Nordisk Investigational Site, Rockville, Maryland
  - Novo Nordisk Investigational Site, Springfield, Massachusetts
  - Novo Nordisk Investigational Site, Buckley, Michigan
  - Novo Nordisk Investigational Site, Southfield, Michigan
  - Novo Nordisk Investigational Site, Great Falls, Montana
  - Novo Nordisk Investigational Site, Nashua, New Hampshire
  - Novo Nordisk Investigational Site, Rosedale, New York
  - Novo Nordisk Investigational Site, Staten Island, New York
  - Novo Nordisk Investigational Site, Greenville, North Carolina
  - Novo Nordisk Investigational Site, Mooresville, North Carolina
  - Novo Nordisk Investigational Site, Franklin, Ohio
  - Novo Nordisk Investigational Site, Mason, Ohio
  - Novo Nordisk Investigational Site, Wadsworth, Ohio
  - Novo Nordisk Investigational Site, Oklahoma City, Oklahoma
  - Novo Nordisk Investigational Site, McMurray, Pennsylvania
  - Novo Nordisk Investigational Site, Norristown, Pennsylvania
  - Novo Nordisk Investigational Site, Philadelphia, Pennsylvania
  - Novo Nordisk Investigational Site, East Providence, Rhode Island
  - Novo Nordisk Investigational Site, Chattanooga, Tennessee
  - Novo Nordisk Investigational Site, Kingsport, Tennessee
  - Novo Nordisk Investigational Site, Amarillo, Texas
  - Novo Nordisk Investigational Site, Lubbock, Texas
  - Novo Nordisk Investigational Site, Sugar Land, Texas
  - Novo Nordisk Investigational Site, Newport News, Virginia
  - Novo Nordisk Investigational Site, Richmond, Virginia
  - Novo Nordisk Investigational Site, Winchester, Virginia
  - Novo Nordisk Investigational Site, Milwaukee, Wisconsin
- France (5):
  - Novo Nordisk Investigational Site, Brest
  - Novo Nordisk Investigational Site, La Roche-sur-Yon
  - Novo Nordisk Investigational Site, La Rochelle
  - Novo Nordisk Investigational Site, Pointe à Pitre
  - Novo Nordisk Investigational Site, Strasbourg
- Poland (6):
  - Novo Nordisk Investigational Site, Bialystok
  - Novo Nordisk Investigational Site, Gdansk
  - Novo Nordisk Investigational Site, Katowice
  - Novo Nordisk Investigational Site, Krakow
  - Novo Nordisk Investigational Site, Poznan
  - Novo Nordisk Investigational Site, Zabrze
- Russia (11):
  - Novo Nordisk Investigational Site, Barnaul
  - Novo Nordisk Investigational Site, Kazan'
  - Novo Nordisk Investigational Site, Kursk
  - Novo Nordisk Investigational Site, Moscow
  - Novo Nordisk Investigational Site, Nizhny Novgorod
  - Novo Nordisk Investigational Site, Penza
  - Novo Nordisk Investigational Site, Saint Petersburg
  - Novo Nordisk Investigational Site, Samara
  - Novo Nordisk Investigational Site, Saratov
  - Novo Nordisk Investigational Site, Smolensk
  - Novo Nordisk Investigational Site, Volgograd
- Ukraine (5):
  - Novo Nordisk Investigational Site, Kharkiv
  - Novo Nordisk Investigational Site, Kiev
  - Novo Nordisk Investigational Site, Kyiv
  - Novo Nordisk Investigational Site, Vinnytsia
  - Novo Nordisk Investigational Site, Zaporizhia
- United Kingdom (8):
  - Novo Nordisk Investigational Site, Bristol
  - Novo Nordisk Investigational Site, Dundee
  - Novo Nordisk Investigational Site, Edinburgh
  - Novo Nordisk Investigational Site, Hull
  - Novo Nordisk Investigational Site, Leicester
  - Novo Nordisk Investigational Site, Letchworth Garden City
  - Novo Nordisk Investigational Site, London
  - Novo Nordisk Investigational Site, Swansea

REFERENCES:
- [Result] Davies MJ, Bain SC, Atkin SL, Rossing P, Scott D, Shamkhalova MS, Bosch-Traberg H, Syren A, Umpierrez GE. Efficacy and Safety of Liraglutide Versus Placebo as Add-on to Glucose-Lowering Therapy in Patients With Type 2 Diabetes and Moderate Renal Impairment (LIRA-RENAL): A Randomized Clinical Trial. Diabetes Care. 2016 Feb;39(2):222-30. doi: 10.2337/dc14-2883. Epub 2015 Dec 17. PMID 26681713
- [Result] Zobel EH, von Scholten BJ, Goldman B, Persson F, Hansen TW, Rossing P. Pleiotropic effects of liraglutide in patients with type 2 diabetes and moderate renal impairment: Individual effects of treatment. Diabetes Obes Metab. 2019 May;21(5):1261-1265. doi: 10.1111/dom.13638. Epub 2019 Feb 22. PMID 30663196
- [Derived] Natale P, Green SC, Tunnicliffe DJ, Pellegrino G, Toyama T, Strippoli GF. Glucagon-like peptide 1 (GLP-1) receptor agonists for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2025 Feb 18;2(2):CD015849. doi: 10.1002/14651858.CD015849.pub2. PMID 39963952
- [Derived] Kim JD, Park CY, Cha BY, Ahn KJ, Kim IJ, Park KS, Lee HW, Min KW, Won JC, Chung MY, Kim JT, Kang JG, Park SW. Comparison of Adherence to Glimepiride/Metformin Sustained Release Once-daily Versus Glimepiride/Metformin Immediate Release BID Fixed-combination Therapy Using the Medication Event Monitoring System in Patients With Type 2 Diabetes. Clin Ther. 2018 May;40(5):752-761.e2. doi: 10.1016/j.clinthera.2018.04.002. Epub 2018 May 3. PMID 29729957
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was conducted in France, Poland, Russian Federation, Ukraine, United Kingdom, and the United States of America.
Groups:
- Lira 1.8 mg: Subjects received subcutaneous (s.c) liraglutide 1.8 mg once daily, applying a 3-4 week dose escalation regimen with weekly increments of 0.6 mg until the maintenance dose of 1.8 mg was reached, as an add-on to the subject's stable pre-trial oral antidiabetic drug (OAD) and/or insulin regimen (monotherapy or any duo-combinations of metformin and/or sulphonylureas and/or pioglitazone; or monotherapy of basal or premix insulin or combination with metformin and/or pioglitazone).
- Placebo: Subjects received s.c placebo 1.8 mg once daily, applying a 3-4 week dose escalation regimen with weekly increments of 0.6 mg until the maintenance dose of 1.8 mg was reached, as an add-on to the subject's stable pre-trial OAD and/or insulin regimen (monotherapy or any duo-combinations of metformin and/or sulphonylureas and/or pioglitazone; or monotherapy of basal or premix insulin or combination with metformin and/or pioglitazone).
Period: Overall Study
Arm/Group | Lira 1.8 mg | Placebo
Started | 140 | 139
Exposed | 140 | 137 (2 subjects did not take trial product)
Completed | 105 | 105 (2 subjects did not take trial product)
Not Completed | 35 | 34
Not completed — Adverse Event | 17 | 4
Not completed — Protocol Violation | 0 | 3
Not completed — Withdrawal Criteria | 17 | 25
Not completed — Unclassified | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lira 1.8 mg | Placebo | Total
Number analyzed (Participants) | 140 | 137 | 277
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.0 (8.3) | 66.3 (8.0) | 67.2 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 72 | 137
  Male | 75 | 65 | 140
Fasting plasma glucose (FPG) [Mean (Standard Deviation); unit: mmol/L] | 9.48 (3.270) | 9.27 (2.842) | 9.38 (3.061)
Glycosylated haemoglobin (%)(HbA1c) [Mean (Standard Deviation); unit: Percent (%) glycosylated haemoglobin] | 8.08 (0.792) | 8.00 (0.853) | 8.04 (0.823)

OUTCOME MEASURES:

1. Primary Outcome: Estimated Mean From the Statistical Model and Standard Deviation From Observed Data For Change From Baseline to Week 26 in HbA1c (%) (Glycosylated Haemoglobin)
Description: Calculated as the estimated mean change from baseline in HbA1c (%) after 26 Weeks of treatment based on the statistical model.
Time Frame: Week 0, Week 26
Population: The full analysis set (FAS) included all randomised subjects that received at least one dose of the study medication. A total of 14 subjects in the FAS did not contribute to the analysis due to missing data.
Measure: Mean (Standard Deviation); unit: percentage (%)
Arm/Group | Lira 1.8 mg | Placebo
Number analyzed (Participants) | 127 | 136
percentage (%) | -1.05 (0.8944) | -0.38 (0.8797)
Statistical Analysis 1: Comparison: Lira 1.8 mg vs Placebo; The null hypothesis of no treatment difference was tested using a two-sided test based on a mixed model repeated measurement (MMRM) analysis. The model included treatment, country, stratification groups (6 groups from cross-classifying renal function category (2 levels: eGFR<45 and ≥45 mL/min) and the background insulin treatment category (3 levels: basal, premix or no insulin)) as fixed effects factors and baseline HbA1c as a covariate, all nested within week; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Adjustment for multiple comparisons was not used since there was only one primary endpoint; Estimated treatment difference = -0.66, 95% CI [-0.90 to -0.43]

2. Secondary Outcome: Estimated Proportion of Responders Achieving HbA1c <7.0% and no Weight Gain After 26 Weeks of Treatment
Description: Calculated as estimated percentage of subjects achieving HbA1c <7.0% and no weight gain after 26 weeks of treatment based on the statistical model.
Time Frame: At week 26
Population: The FAS included all randomised subjects that received at least one dose of study medication. A total of 14 subjects in the FAS did not contribute to the analysis due to missing data.
Measure: Number; unit: percentage of patients
Arm/Group | Lira 1.8 mg | Placebo
Number analyzed (Participants) | 127 | 136
percentage of patients | 46.03 | 15.99
Statistical Analysis 1: Comparison: Lira 1.8 mg vs Placebo; Analysed by a logistic regression model with treatment, country and stratification groups as fixed effects and HbA1c and body weight at baseline as covariates. No weight gain was defined as change from baseline to Week 26 in body weight ≤0 kg; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Not adjusted for multiple comparisons; Estimated odds ratio = 4.48, 95% CI [2.46 to 8.18]

3. Secondary Outcome: Estimated Proportion of Responders Achieving HbA1c <7.0% and no Minor or Severe Hypoglycaemic Episodes After 26 Weeks of Treatment
Description: Calculated as estimated percentage of subjects achieving HbA1c <7.0% and no minor or severe hypoglycaemic episodes observed within 26 weeks of treatment based on the statistical model.
Time Frame: At week 26
Population: as for outcome 2
Measure: Number; unit: percentage of patients
Arm/Group | Lira 1.8 mg | Placebo
Number analyzed (Participants) | 127 | 136
percentage of patients | 33.23 | 11.23
Statistical Analysis 1: Comparison: Lira 1.8 mg vs Placebo; Analysed by a logistic regression model with treatment, country and stratification groups as fixed effects and HbA1c at baseline as covariates; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Not adjusted for multiple comparisons; Estimated odds ratio = 3.94, 95% CI [2.12 to 7.30]

4. Secondary Outcome: Estimated Mean From the Statistical Model and Standard Deviation From Observed Data For Change From Baseline to Week 26 in Self-measured Plasma Glucose (SMPG) 7-point Profiles
Description: SMPG was measured before and 90 minutes after breakfast, lunch and dinner and at bedtime at Week 0, 12 and 26. A summary measure of the 7 values was derived for each applicable visit as the area under the curve divided by the period of time elapsed between the first and last measurement. The change from baseline to week 26 was estimated using the statistical model.
Time Frame: Week 0, week 26
Population: The FAS included all randomised subjects that received at least one dose of study medication. A total of 46 subjects in the FAS did not contribute to the analysis due to missing data.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Lira 1.8 mg | Placebo
Number analyzed (Participants) | 109 | 122
mmol/L | -1.59 (2.480) | -0.51 (2.391)
Statistical Analysis 1: Comparison: Lira 1.8 mg vs Placebo; Mean change from baseline in the 7-point profile (SMPG) after 26 weeks treatment was analysed using an MMRM model with treatment, country and stratification groups as fixed effects and baseline as a covariate, all nested within visit; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Not adjusted for multiple comparisons; Estimated treatment difference = -1.08, 95% CI [-1.58 to -0.58]

5. Secondary Outcome: Estimated Mean From the Statistical Model and Standard Deviation From Observed Data For Change From Baseline to Week 26 in Body Mass Index (BMI)
Description: Calculated as estimated mean change in BMI (kg/m˄2) from baseline to Week 26 based on the statistical model.
Time Frame: Week 0, week 26
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Lira 1.8 mg | Placebo
Number analyzed (Participants) | 127 | 136
kg/m^2 | -0.88 (1.3214) | -0.38 (1.1679)
Statistical Analysis 1: Comparison: Lira 1.8 mg vs Placebo; Change from baseline in BMI (kg/m˄2) after 26 weeks treatment was analysed separately using an MMRM analysis model with treatment, country and stratification groups as fixed effects and baseline as a covariate, all nested within visit; Test type: Superiority or Other; p = 0.0022, Mixed Models Analysis; Not adjusted for multiple comparisons; Estimated treatment difference = -0.51, 95% CI [-0.83 to -0.18]

6. Secondary Outcome: Estimated Mean Ratio to Baseline and Observed Coefficient of Variation in Renal Function-estimated Glomerular Filtration Rate (eGFR) (to Check How Well the Kidneys Are Functioning Using Modification of Diet in Renal Disease (MDRD) Formula)
Description: Calculated as the estimated ratio to baseline in eGFR (mL/min/1.73m˄2) after 26 Weeks of treatment based on the statistical model.
Time Frame: Week 0, week 26
Population: Safety analysis set included all subjects receiving at least one dose of the trial product. A total of 8 subjects in the safety analysis set did not contribute to the analysis due to missing data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min/1.73m˄2
Arm/Group | Lira 1.8 mg | Placebo
Number analyzed (Participants) | 132 | 137
mL/min/1.73m˄2 | 0.99 (0.17) | 1.01 (0.19)
Statistical Analysis 1: Comparison: Lira 1.8 mg vs Placebo; The ratio to baseline in eGFR (mL/min/1.73m˄2) after 26 weeks treatment was estimated based on log-transformed data for changes from baseline. The responses were analysed using an MMRM model with treatment, country and stratification groups as fixed effects and log-transformed baseline as a covariate, all nested within visit. The resulting estimates were back-transformed to the original scale; Test type: Superiority or Other; p = 0.3575, Mixed Models Analysis — Not adjusted for multiple comparisons; Estimated treatment ratio = 0.98, 95% CI [0.94 to 1.02]

ADVERSE EVENTS:
Time Frame: The adverse events were collected from Week 0 to Week 27±3 Days
Description: Safety analysis set included all subjects receiving at least one dose of the investigational product.
Arm/Group | Lira 1.8 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 14/140 | 15/137
Other Adverse Events (participants affected / at risk) | 73/140 | 49/137
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lira 1.8 mg (N=140) | Placebo (N=137)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
Autoimmune hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Arteriosclerotic gangrene (Infections and infestations) | 0 (0) | 1 (1)
Biliary sepsis (Infections and infestations) | 1 (1) | 0 (0)
Meningitis herpes (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal cord injury lumbar (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0)
Glomerular filtration rate decreased (Investigations) | 0 (0) | 1 (1)
Urine albumin/creatinine ratio increased (Investigations) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign neoplasm of cervix uteri (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (1) | 1 (1)
Urethral stenosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Colectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1)
Poor peripheral circulation (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lira 1.8 mg (N=140) | Placebo (N=137)
Constipation (Gastrointestinal disorders) | 8 (9) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 10 (13) | 4 (6)
Nausea (Gastrointestinal disorders) | 30 (39) | 6 (10)
Vomiting (Gastrointestinal disorders) | 17 (18) | 3 (4)
Nasopharyngitis (Infections and infestations) | 7 (7) | 16 (17)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 7 (8)
Glomerular filtration rate decreased (Investigations) | 9 (10) | 7 (14)
Lipase increased (Investigations) | 21 (23) | 12 (13)
Headache (Nervous system disorders) | 7 (8) | 4 (8)
Renal impairment (Renal and urinary disorders) | 7 (7) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk maintains the right to be informed of any Investigator plans for publication and to review any scientific paper, presentation, communication or other information concerning the investigation described in this protocol. Any such communication must be submitted in writing to the Novo Nordisk trial manager prior to submission for comments. Comments will be given within four weeks from receipt of the planned communication.